CLINICAL TRIAL: NCT03452605
Title: Effect of Acute Cocoa Flavanol Intake on the BOLD Response and Cognitive Function in Patients With Type 1 Diabetes
Brief Title: The Effect of Cocoa Flavanol on the BOLD Response and Cognitive Function in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Prof., Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: T1DCFMRI
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high cocoa flavanol drink (Experimental): high cocoa flavanol drink (900 mg cocoa flavanol dissolved in 300 ml skimmed milk) 2h pre-fMRI
  Interventions: Dietary Supplement: cocoa flavanol supplementation
- low cocoa flavanol drink (Placebo Comparator): low cocoa flavanol drink (30 mg cocoa flavanol dissolved in 300 ml skimmed milk), matched for theobromine, caffeine and macronutrients with the high cocoa flavanol drink 2h-pre fMRI
  Interventions: Dietary Supplement: cocoa flavanol supplementation

INTERVENTIONS:
Dietary Supplement: cocoa flavanol supplementation — cocoa flavanols (containing 196 mg epicatechin)

SUMMARY:
Type 1 Diabetes (T1D) is associated with microvascular changes in the brain, which can cause cognitive dysfunction. Cocoa flavanols (CF) can stimulate vasodilation, resulting in enhanced cerebral blood flow and better cognitive function. This study aimed to investigate whether acute CF supplementation can improve cognitive function and the hemodynamic (BOLD) response in T1D patients.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking T1D patients or matched healthy controls
* having diabetes for more than 1 year
* males and females older than 18 years
* stable medications for more than 6 months (no use of cholinesterase inhibitors or prior use of multivitamins was allowed)
* adequate visual and auditory acuity to allow neuropsychological testing.

Exclusion Criteria:

* participant enrolled in any investigational drug study within 2 months or longer, depending on the investigational drug half-life
* history in the past 2 years of epileptic seizures or any major psychiatric disorder
* history or MRI evidence of brain damage, including significant trauma, stroke, hydrocephalus, mental retardation, or serious neurological disorder,
* significant history of alcoholism or drug abuse
* unstable cardiac, renal, lung, liver, or other severe chronic disease
* hypertension (systolic blood pressure ≥160 mmHg, diastolic blood pres-sure ≥100 mmHg) or hypotension (systolic blood pressure <100 mmHg)
* pacemaker or other medical metal devices that precludes performing MRI,
* chronic inflammatory diseases, including lupus, rheumatoid arthritis, or polymyalgia rheumatic
* macrovascular complications
* retinopathy, nephropathy or neuropathy (microvascular complications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
cognitive function | 5 min
  reaction time (milliseconds) on the flanker task
BOLD fmri response | 5 min
  blood oxygenation level dependent response during flanker test